CLINICAL TRIAL: NCT07390838
Title: An Open, Multicenter, Phase I Clinical Study on the Safety, Efficacy, and Pharmacokinetics of SH009 Injection in Patients With Advanced Solid Tumors.
Brief Title: A Study of SH009 Injection in Patients With Advanced Solid Tumors.
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Nanjing Sanhome Pharmaceutical, Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SHS009-I-03
Record Dates: First submitted 2026-01-13; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Liver Cancer (Locally Advanced or Metastatic); Lung Cancer (NSCLC); Head and Neck Cancer Squamous Cell Carcinoma; Breast Cancer (Locally Advanced or Metastatic); Esophageal Cancer; Gastric Cancer (GC); Solid Tumor Malignancies
MeSH Terms: conditions — Liver Neoplasms; Neoplasm Metastasis; Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Breast Neoplasms; Esophageal Neoplasms; Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SH009 (Experimental)
  Interventions: Drug: SH009

INTERVENTIONS:
Drug: SH009 — The dosage of SH009 is 40 mg/kg QW with a treatment cycle of 28 days

SUMMARY:
Evaluate the efficacy and safety of SH009 injection therapy for patients with advanced solid tumors

DETAILED DESCRIPTION:
Based on the obtained data from the dose escalation phase of the Phase I clinical trial, select safe and effective tumor indications (including but not limited to gastric cancer, liver cancer, head and neck tumors, breast cancer, non-small cell lung cancer, esophageal cancer, etc.) and dose levels for dose expansion studies. Further evaluate efficacy, safety, and pharmacokinetics to provide a basis for determining the recommended dose for Phase II clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* (1) Age≥18 years old at the time of informed consent, male or female;
* (2) Subjects with histologically confirmed locally advanced, recurrent, or metastatic solid tumors (including but not limited to colorectal cancer, gastric cancer, hepatocellular carcinoma, head and neck cancer, breast cancer, non-small cell lung cancer, esophageal cancer, etc.) who have experienced disease progression or intolerance to at least one prior line of systemic therapy, and for whom no acceptable standard therapy exists or who cannot benefit from or tolerate standard therapy;
* (3) Subjects must have at least one measurable lesion per RECIST 1.1 criteria. A lesion that has been previously irradiated can only be considered measurable if there is documented progression at that site following radiotherapy;
* (4) Archival tumor tissue samples are available, or the subject agrees to undergo a tumor biopsy for the determination of PD-L1 and CD47 expression levels and other biomarker analyses;
* (5) Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 to 2;
* (6) Life expectancy ≥12 weeks;
* (7) Bone marrow function meets the following criteria: neutrophil count ≥ 1.5 × 10^9/L; platelet count ≥ 90 × 10^9/L (platelet count ≥ 75 × 10^9/L in patients with liver cancer); hemoglobin (Hb) ≥ 90 g/L;
* (8) Liver function meets the following criteria: total bilirubin(TBIL) ≤ 1.5 × ULN (total bilirubin ≤ 3 × ULN for subjects with Gilbert's syndrome); aspartate aminotransferase (AST) and alanine and aminotransferase (ALT) ≤ 3 × ULN (ALT and AST ≤ 5 × ULN for subjects with liver cancer or liver metastases);
* (9) Renal function meets the following criteria: serum creatinine clearance(CLcr) ≥ 50 mL/min (calculated according to Cockcroft-Gault formula); urine dipstick test results show that urine protein < 2 +, urine protein ≥ 2 + subjects should undergo 24-hour urine collection and urine protein content < 1g within 24 hours;
* (10) Coagulation function meets the following criteria: prothrombin time (PT), activated partial thromboplastin time (APTT) and international normalized ratio (INR) ≤ 1.5× ULN;
* (11) Female subjects of childbearing potential must use effective contraception during the trial and for 6 months after the last dose, and have a negative pregnancy test within 7 days before treatment initiation (except those who are surgically sterilized or postmenopausal). Male subjects must agree to use effective contraception during the trial and for 6 months after the last dose;
* (12) The subject is fully informed about this trial before its commencement and voluntarily signs and dates the informed consent form.

Exclusion Criteria:

* (1) Prior exposure to any CD47 antibody, SIRPα antibody, or CD47/SIRPα recombinant protein;
* (2) Prior treatment with adoptive cellular therapies such as CAR-T, TCR-T, or TIL. Prior administration of an anti-cancer vaccine, or use of live or live-attenuated vaccines within 4 weeks prior to the first dose;
* (3) Systemic anti-tumor therapies within the specified timeframes prior to the first dose of study drug: Chemotherapy, antibody-based targeted therapy, endocrine therapy, or immunotherapy within 3 weeks. Mitomycin or nitrosoureas within 6 weeks. Oral fluoropyrimidines (e.g., S-1, capecitabine) and small molecule targeted agents within 2 weeks or 5 half-lives of the drug (whichever is longer).Chinese/herbal medicines with anti-cancer activity indicated in their labeling must be discontinued prior to enrollment. Prior radical radiotherapy within 3 months before study drug administration is excluded. Palliative radiotherapy administered within 2 weeks prior to dosing is allowed if the dose meets local palliative care standards and the radiation field covers less than 30% of the bone marrow area;
* (4) Received any investigational drug within 28 days before administration of this trial, or participated in another clinical study at the same time, except for the following circumstances: the patient participated in an observational, non-interventional clinical study, or was in the follow-up period after the end of treatment in an interventional clinical study but the drug withdrawal had exceeded the washout period;
* (5) Had major organ surgery (excluding puncture biopsy) or had significant trauma within 4 weeks before the first administration, or needed to undergo elective surgery during the trial period;
* (6) Patients who received systemic glucocorticoids (dexamethasone > 10 mg/ day or equivalent dose of the same drug) or other immunosuppressive therapy within 14 days before the first administration; except for topical, ocular, intra-articular, intranasal, and inhaled glucocorticoids; short-term use of glucocorticoids for prophylactic treatment (e.g., prevention of contrast allergy);
* (7) Symptomatic brain parenchymal or leptomeningeal metastases, deemed by the investigator as unsuitable for enrollment;
* (8) Prior immunotherapy with ≥Grade 3 irAE or ≥Grade 2 immune-related myocarditis;
* (9) Severe or uncontrolled systemic disease, including but not limited to: uncontrolled pleural or peritoneal effusion; uncontrolled diabetes; ventricular arrhythmia requiring intervention; acute coronary syndrome, congestive heart failure, stroke, or other ≥Grade 3 cardiovascular event within 6 months; NYHA Class ≥II or LVEF <50%; clinically significant QTcF prolongation or arrhythmia risk (baseline QTcF >450 msec for males or >470 msec for females); clinically uncontrolled hypertension (SBP >160 mmHg and/or DBP >90 mmHg after treatment) as judged by the investigator. Subjects judged by the investigator as unsuitable due to any such condition;
* (10) History of pneumonia requiring hormone therapy or interstitial lung disease (including past and current history); active pulmonary infection;
* (11) Active infection requiring intravenous anti-infective therapy within 1 week prior to study drug administration (fever attributed to the tumor per investigator's judgment is acceptable). History of self-limited infections that have resolved is acceptable;
* (12) Active Hepatitis B, Hepatitis C, or syphilis infection. Subjects positive for HBeAb or HBsAg are eligible if HBV-DNA ≤200 IU/mL. Subjects positive for HCV-Ab are eligible if HCV-RNA ≤ the upper limit of normal at the research center. Subjects with hepatocellular carcinoma and HBV-DNA ≥2000 IU/mL must receive antiviral/hepatoprotective therapy first and can only enroll after HBV-DNA decreases to <2000 IU/mL;
* (13) History of primary immunodeficiency, including positive human immunodeficiency virus (HIV) test, or suffering from other acquired, congenital immunodeficiency diseases;
* (14) History of other malignancies within 5 years prior to the first dose, except for:

  a) Any other invasive malignancy, treated with curative intent, with a disease-free interval >3 years and deemed by the investigator not to affect efficacy evaluation for the current tumor. b) Adequately treated basal cell or squamous cell skin cancer, superficial bladder cancer, carcinoma in situ of the cervix or breast, or other locally cured cancers;
* (15) History or presence of autoimmune disease within 2 years, including but not limited to systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, autoimmune thyroid disease, multiple sclerosis, vasculitis, glomerulonephritis or high risk (e.g., post-transplant immunosuppression). Exceptions: stable type 1 diabetes on fixed-dose insulin; autoimmune hypothyroidism on hormone replacement only; skin conditions not requiring systemic treatment (e.g., eczema, rash covering<10% BSA, psoriasis without ocular symptoms);
* (16) Arterial thromboembolic events within 6 months prior to the first dose, including myocardial infarction, unstable angina, cerebrovascular accident, or transient ischemic attack. History of deep vein thrombosis, pulmonary embolism, or other serious thromboembolism within 3 months prior to the first dose (catheter-related or superficial venous thrombosis is not considered "serious"). Receiving thrombolytic or anticoagulant therapy for high thrombotic risk;
* (17) Subjects who had receive allogeneic hematopoietic stem cell transplantation or solid organ transplantation (except corneal transplant);
* (18) According to CTCAE 5.0, adverse reactions from previous anti-tumor therapy have not yet returned to ≤ grade 1 (except for toxicities which are judged by researchers to be safe, such as hair loss, pigmentation, hypothyroidism stabilized by hormone replacement therapy and peripheral neuropathy (need to recover to ≤ grade 2)). Irreversible toxicity (e.g., hearing loss) that is not reasonably expected to be aggravated by the study drug may be allowed after consultation with the medical monitor;
* (19) Known history of severe hypersensitivity to macromolecular protein preparations/monoclonal antibodies(CTCAE v5.0 Grade ≥3), or any component of the study drug;
* (20) Known alcohol and/or drug dependence, or any other condition deemed by the investigator to affect the safety or compliance of the study treatment, including but not limited to psychiatric disorders;
* (21) Pregnant or lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-05-16 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | up to 2 years
  Proportion of subjects who have a complete or partial response as assessed according to RECIST v1.1
Duration of response (DoR) | up to 2 years
  Duration of response (DoR), which is defined as the duration from the first documentation of objective response to the first documented disease progression or death due to any cause, whichever occurs first
Time to response (TTR) | up to 2 years
  TTR is defined as the time to response base on RECIST v1.1
Disease control rate (DCR) | up to 2 years
  Disease control rate (DCR), which is defined as the proportion of subjects with complete response (CR), partial response (PR), or stable disease (SD), based on RECIST v1.1
Progression-free survival (PFS) | up to 2 years
  From date of enrollment until the date of first documented progression or date of death from any cause, whichever came first
Overall survival (OS) | up to 2 years
  From date of enrollment until the date of death from any cause

SECONDARY OUTCOMES:
Percentage of participants with adverse event (AE) | From the subject signs the Informed Consent Form to 30 days (AE) and 90 days (Serious AE) after the last dose of study treatment or initiation of other anti-tumor therapy, whichever occurs first,up to 2 years
  The percentage of participants experiencing an adverse event (AE) and the severity of AEs will be assessed
Observed concentrations of SH009 | From date of enrollment until the end of treatment, assessed up to 2 years
  The endpoints for assessment of Pharmacokinetics (PK) of SH009 include serum concentrations of SH009 at different timepoints after SH009 administration
Number of participants who develop detectable anti-drug antibodies (ADAs) | From first dose of SH009 through 90 days after last dose of SH009, up to 2 years
  The immunogenicity of SH009 will be assessed by summarizing the number of participants who develop detectable antidrug antibodies (ADAs)

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Gaobo Cancer Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No